CLINICAL TRIAL: NCT05577468
Title: A Multi-center, Randomized, Double-blind, Double-dummy Phase III Clinical Study to Evaluate the Efficacy and Safety of Tegoprazan Versus Esomeprazole-containing Bismuth Quadruple Therapy for Eradication of Helicobacter Pylori
Brief Title: Efficacy and Safety of Tegoprazan Versus Esomeprazole-containing Bismuth Quadruple Therapy for Eradication of Helicobacter Pylori
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shandong Luoxin Pharmaceutical Group Stock Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NC822101
Record Dates: First submitted 2022-10-09; First posted 2022-10-13 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — tegoprazan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tegoprazan (Experimental): Participants will receive Tegoprazan tablets Esomeprazole magnesium enteric-coated tablets placebo Bismuth potassium citrate capsules Amoxicillin capsules Clarithromycin tablets
  Interventions: Drug: Tegoprazan
- Esomeprazole (Active Comparator): Participants will receive Tegoprazan tablets placebo Esomeprazole magnesium enteric-coated tablets Bismuth potassium citrate capsules Amoxicillin capsules Clarithromycin tablets
  Interventions: Drug: Tegoprazan

INTERVENTIONS:
Drug: Tegoprazan — tegoprazan-containing bismuth quadruple therapy or Esomeprazole-containing bismuth quadruple therapy; Route of administration: oral;

SUMMARY:
This study is a multicenter, randomized, double-blind, double-dummy, phase III study to evaluate the efficacy and safety of tegoprazan versus esomeprazole-containing bismuth quadruple therapy in patients infected with Helicobacter pylori in China.

Screening phase: After signing the informed consent form, subjects will be determined for Helicobacter pylori infection by 13^C-urea breath test (UBT),histological testing and bacterial culture during the screening period. Subjects who meet all screening criteria will be randomized in a 1:1 ratio to receive the tegoprazan-containing bismuth quadruple therapy (hereinafter referred to as the tegoprazan group) or esomeprazole-containing bismuth quadruple therapy (hereinafter referred to as the esomeprazole group).

Treatment phase: Subjects will receive relevant study medication starting on Day 1 of the treatment period for 14 days.

Follow-up phase: Within 29+7 days after the last study drug treatment, subjects will return to the study site for efficacy and safety assessments. 13^C-UBT detection will be performed in this follow-up visit to determine the Hp infection status of the subjects after treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1) Subjects who volunteer to sign the written informed consent form approved by the Ethics Committee and agree to participate in this study prior to the initiation of any study procedures.

  2) Subjects who are able to understand and follow the protocol requirements and agree to participate in all the study visits.

  3) Males or females ≥18 years old and ≤70 years old. 4) In the screening stage, subjects are confirmed Hp infection by 13^C-urea breath test , histology test and bacterial culture, and then the investigators judge that Hp eradication treatment is required.

  5) Subjects who agree to use appropriate medical method for contraception during the course of the study (not including women in medically sterile state)

Exclusion Criteria:

* 1) Subjects received Hp eradication treatment previously. 2) Subjects who have participated in other clinical studies within 4 weeks before screening, except for the following two situations:
* The study which the subject is participating or participated in is a non-interventional study (e.g. observational study or questionnaire survey); Subject had signed the informed consent form in that study, but withdrew from that study prior to the start of any treatment.
* Subjects who have participated in the [NC821604] study and have demonstrated ulcer healing may participate in this study.

  3) Subjects who participated in the planning and execution of this study. 4) Women who are pregnant or breastfeeding. 5) Subjects with known allergy to tegoprazan, esomeprazole, penicillins or other β-lactams, macrolide antibiotics or bismuth (including any related excipients). If a skin sensitivity test (skin test) is required, it should be carried out at Visit 1 according to routine medical practice.

  6) Subjects with a history of drug (including but not limited to opioids) abuse or alcohol abuse within 1 year before the screening visit.

  7) Subjects with Zollinger-Ellison syndrome. 8) Subjects who have previously undergone surgery or operations that may affect gastric acid secretion or drug absorption, 9) Subjects with "warning" symptoms such as painful swallowing, severe dysphagia, bleeding, weight loss, anemia, or blood in the stool that may indicate malignant lesions of the gastrointestinal tract, unless the possibility of malignant lesions is ruled out by endoscopy.

  10) Subjects with a history of malignant tumor within 5 years before screening 11) Subjects who cannot undergo upper gastrointestinal endoscopy. 12) Subjects whose upper gastrointestinal endoscopy demonstrates acute upper gastrointestinal bleeding, active gastric ulcer or duodenal ulcer, acute gastric mucosal injury or duodenal mucosal injury.

  13) Subjects with uncontrolled and unstable hepatic, renal, cardiovascular, respiratory, gastrointestinal, endocrine, hematologic, central nervous system or mental diseases as judged by investigators, in which participation in the study may affect the interpretation of their safety or research results.

  14) Subjects who plan to be hospitalized for surgical treatment during the study.

  15) Subjects who have taken H2 receptor antagonists or PPI within 14 days before the 13C-urea breath test during the screening period, or those who have taken antibacterial drugs, bismuth and certain Chinese medicines with antibacterial effects within 28 days before the 13C-urea breath test during the screening period.

  16) Subjects who need to use the prohibited drugs listed in the protocol. 17) Subjects with any of the following laboratory test abnormalities at screening:
* AST > upper limit of normal (ULN);
* ALT > ULN;
* Total bilirubin > 1.2 × ULN;
* Creatinine > 1.5 × ULN; 18) Subjects with clinically significant electrocardiogram (ECG) abnormalities at the screening as judged by investigators.

  19) Human immunodeficiency virus (HIV) antibody positive, hepatitis B virus (HBV) surface antigen positive or hepatitis C virus (HCV) antibody positive confirmed by tests.

  20) Judged by the investigator, there are other conditions compromising the subject's eligibility for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2022-10-30 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of All Participants With Successful Helicobacter Pylori (H.Pylori) Eradication | Day 29+7 days following the completion of treatment(duration of treatment was 2 weeks)
  Percentage of all patients with Hp eradication determined by a 13^C-urea breath test after study treatment.

SECONDARY OUTCOMES:
Percentage of Participants With Successful Helicobacter Pylori (H.Pylori) Eradication in Participants With a Clarithromycin-resistant Strain of H Pylori at Baseline | Day 29+7 days following the completion of treatment( duration of treatment was 2 weeks)
Percentage of Participants With Successful Helicobacter Pylori (H.Pylori) Eradication in Participants With a Clarithromycin-sensitive Strain of H Pylori at Baseline | Day 29+7 days following the completion of treatment(duration of treatment was 2 weeks)
Percentage of Participants With Successful Helicobacter Pylori (H.Pylori) Eradication in Participants With a Amoxicillin-resistant Strain of H Pylori at Baseline | Day 29+7 days following the completion of treatment(duration of treatment was 2 weeks)
Percentage of Participants With Successful Helicobacter Pylori (H.Pylori) Eradication in Participants With a Amoxicillin-sensitive Strain of H Pylori at Baseline | Day 29+7 days following the completion of treatment(duration of treatment was 2 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Song Z, Wang W, Li P, Zuo X, Zhu Y, Chen Y, Zhang X, Lyu B, Lin R, Du Y, Lan C, Wu H, Chen W, Ye Y, Fan H, Liao A, Chen H, Liu C, Zhang Z, Wang W, Suo Z, Li X, Du Q, Li X, Pan F, Tang J, Xu M, Liu X, Zheng P, Chen H, Du L, Lu J, Feng C, Pan W, Wang H, Zeng Z, Wang J, Lyu S, Liu D, Yang S, Li L, Zhou L. Tegoprazan-based versus esomeprazole-based triple therapy plus bismuth for first-line Helicobacter pylori eradication: A nationwide, multicenter, double-blind, double-dummy, randomized controlled trial. Chin Med J (Engl). 2025 Aug 22. doi: 10.1097/CM9.0000000000003780. Online ahead of print. PMID 40846665